CLINICAL TRIAL: NCT01421576
Title: A Randomized, Single-dose, 2-sequence, 2-period Crossover Study to Investigate the Food-effect Pharmacokinetics of Sarpogrelate HCl Controlled Release Tablet in Healthy Male Subjects
Brief Title: Bioavailability Study of DP-R202 in Healthy Male Volunteers Under Fed Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Alvogen Korea (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: DP-SACL-I-002
Record Dates: First submitted 2011-08-09; First posted 2011-08-23 (Estimated); Last update posted 2011-08-23 (Estimated); Status verified 2011-08

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- High fat meal (Active Comparator)
  Interventions: Dietary Supplement: High fat meal
- DP-R202 (Experimental): under fed condition
  Interventions: Dietary Supplement: High fat meal

INTERVENTIONS:
Dietary Supplement: High fat meal — offer high fat-meal in the morning before drug intake.
  Other Names: Other Names:; DP-R202 : DP11002-3

SUMMARY:
A randomized, open-label, single-dose, crossover clinical trial to evaluate the food effect on the pharmacokinetics of DP-R202 tablet after oral administration in healthy male volunteers.

DETAILED DESCRIPTION:
The number of patient is twenty-four.Patients were randomly assigned either DP-R202(Sarpogrelate HCL 300mg, qd) under fasting condition or DP-R202(Sarpogrelate HCL 300mg, qd) after eating foods.

ELIGIBILITY:
Inclusion Criteria:

* 20 to 55 years of healthy volunteers

Exclusion Criteria:

* Hypersensitivity Reaction about Sarpogrelate HCL or other antiplatelets

Ages: 20 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2011-07; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Composite of Pharmacokinetics(Cmax, AUClast) | 24h

CONTACTS AND LOCATIONS:
Overall Officials: Jae Wook Ko, M.D., Ph.D, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, Gangnam, South Korea